CLINICAL TRIAL: NCT00044044
Title: A 6-Week, Double-Blind, Randomized, Fixed-Dose, Parallel-Group Study of the Efficacy and Safety of Three Dose Levels of SM-13496 Compared to Placebo and Haloperidol in Patients With Schizophrenia Who Are Experiencing an Acute Exacerbation of Symptoms
Brief Title: A Comparison of Study Drug With Placebo and Haloperidol in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D1050049
Record Dates: First submitted 2002-08-16; First posted 2002-08-20 (Estimated); Results first posted 2011-04-12 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Latuda; Lurasidone
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Lurasidone 20 mg (Experimental): Lurasidone 20 mg tablets
  Interventions: Drug: Lurasidone 20 mg
- Lurasidone 40 mg (Experimental): Lurasidone 40 mg tablets
  Interventions: Drug: Lurasidone 40mg
- Lurasidone 80 mg (Experimental): Lurasidone 2 40 mg tablets
  Interventions: Drug: Lurasidone 80 mg
- Haloperidol 10mg (Active Comparator): Haloperidol 10mg tablets
  Interventions: Drug: Haloperidol 10mg
- Placebo (Placebo Comparator): Matching Placebo to Lurasidone and Haloperidol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lurasidone 20 mg — Lurasidone 20mg/day tablets
  Arms: Lurasidone 20 mg
Drug: Lurasidone 40mg — Lurasidone 40mg/day tablets
  Arms: Lurasidone 40 mg
Drug: Lurasidone 80 mg — Lurasidone 80mg/day - 2 40mg tablets
  Arms: Lurasidone 80 mg
Drug: Haloperidol 10mg — Haloperidol 10mg/day tablets
  Arms: Haloperidol 10mg
Drug: Placebo — Matching Placebo to Lurasdione and Haloperidol
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of the drug SM-13496 compared to a placebo and to haloperidol in patients with schizophrenia.

ELIGIBILITY:
Inclusion criteria:

* The patient has a primary diagnosis of schizophrenia
* The patient has been hospitalized with acute or relapsing schizophrenia within 3 weeks of screening
* The patient has had a duration of illness of at least one year.
* The patient has a BPRS score of at least 42 at baseline and a score of at least 4 in two or more items of the positive symptom subcluster on the PANSS
* The patient is able to remain off antipsychotic medication for a 4 day washout period

Exclusion criteria:

* The patient has had psychiatric hospitalizations other than current hospitalizations within 1 month prior to screening.
* The patient is considered treatment resistant-Substance abuse-Prolactin level of > 200 ng/mL at baseline
* Pregnancy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 356 (Actual)
Dates: Start 2002-07; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (34):
- United States (34):
  - Birmingham Psychiatry Pharmaceutical, Birmingham, Alabama
  - Institute for Psychopharmacology Research, Cerritos, California
  - CNS Network, Garden Grove, California
  - California Clinical Trials Medical Group, Glendale, California
  - Optimum Health Services, La Mesa, California
  - University of California, Irvine, Orange, California
  - Affiliated Research Institute, San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - California Neuropsychopharmacolgoy Clinical Research Insitute, San Diego, California
  - Comprehensive Neuroscience. Inc., Washington D.C., District of Columbia
  - Comprehensive Neuroscience. Inc., Melbourne, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - University of South Florida, Tampa, Florida
  - Coordinated Research of Florida, Inc., Winter Park, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Carman Research, Smyrna, Georgia
  - Hawaii Research Center, Honolulu, Hawaii
  - Alexian Brothers Behavioral Health Hospital, Hoffman Estates, Illinois
  - American Medical Research, Oak Brook, Illinois
  - Centers for Behavioral Health, LLC, Rockville, Maryland
  - Lake Mead Hospital, North Las Vegas, Nevada
  - Comprehensive Clinical Research CNS, PC, Clementon, New Jersey
  - ClinSearch, Inc., Kenilworth, New Jersey
  - Psychiatric Professional Services Inc, Cincinnati, Ohio
  - Quantum Clinical Services Group, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center - Dept. of Psychiatry, Philadelphia, Pennsylvania
  - Community Clinical Research, Austin, Texas
  - FutureSearch Trials, Austin, Texas
  - Claghorn Lesem Research Clinic, Inc., Bellaire, Texas
  - St. Paul Medical Center, Dallas, Texas
  - University Hills Clinical Research, Dallas, Texas
  - CNS, Inc., Falls Church, Virginia
  - Northwest Clinical Research Center, Belleview, Washington
  - Medstream, Inc., Milwaukee, Wisconsin

REFERENCES:
- [Derived] Storman D, Koperny M, Styczen K, Datka W, Jaeschke RR. Lurasidone versus typical antipsychotics for schizophrenia. Cochrane Database Syst Rev. 2025 Jan 20;1(1):CD012429. doi: 10.1002/14651858.CD012429.pub2. PMID 39831535

RESULTS

PARTICIPANT FLOW:
Groups:
- 20 mg: Lurasidone 20 mg oral tablet taken once a day. The number of subjects in the participant flow for the lurasidone 20mg group(overall study) is based on the total number of subjects randomized in this treatment group.
- 40 mg: Lurasidone 40 mg oral tablet taken once a day. The number of subjects in the participant flow for the lurasidone 40mg group(overall study) is based on the total number of subjects randomized in this treatment group.
- 80 mg: Lurasidone 80 mg oral tablet taken once a day. The number of subjects in the participant flow for the lurasidone 80mg group(overall study) is based on the total number of subjects randomized in this treatment group.
- 10 mg Haloperidol: 10 mg Haloperidol overencapsulated tablet taken orally once a day. The number of subjects in the participant flow for the haloperidol 10mg group(overall study) is based on the total number of subjects randomized in this treatment group.
- Placebo: Oral Capsule matching treatment group taken oce a day. The number of subjects in the participant flow for the placebo group(overall study) is based on the total number of subjects randomized in this treatment group.
Period: Overall Study
Arm/Group | 20 mg | 40 mg | 80 mg | 10 mg Haloperidol | Placebo
Started | 71 | 69 | 71 | 73 | 72
Completed | 27 | 28 | 31 | 29 | 36
Not Completed | 44 | 41 | 40 | 44 | 36

BASELINE CHARACTERISTICS:
Groups:
- 20 mg: Lurasidone 20 mg oral tablet taken once a day
- 40 mg: Lurasidone 40 mg oral tablet taken once a day. The number of subjects in the participant flow (overall study) is based on the total number of subjects randomized (356). The number of subjects in the baseline characteristics is based on the safety population (353). All randomized subjects who received at least one dose of study medication were included in the safety analysis. Two subjects who were randomized to the 40 mg treatment group did not take any study medication.
- 80 mg: Lurasidone 80 mg oral tablet taken once a day
- 10 mg Haloperidol: 10 mg Haloperidol overencapsulated tablet taken orally once a day. The number of subjects in the participant flow (overall study) is based on the total number of subjects randomized (356). The number of subjects in the baseline characteristics is based on the safety population (353). All randomized subjects who received at least one dose of study medication were included in the safety analysis. One subject who was randomized to the 10 mg haloperidol treatment group did not take any study medication.
- Placebo: Oral Capsule matching treatment group taken oce a day
- Total: Total of all reporting groups
Arm/Group | 20 mg | 40 mg | 80 mg | 10 mg Haloperidol | Placebo | Total
Number analyzed (Participants) | 71 | 67 | 71 | 72 | 72 | 353
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (10.5) | 42.0 (10.9) | 42.2 (8.3) | 40.0 (10.5) | 41.0 (9.7) | 41.2 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 19 | 14 | 17 | 91
  Male | 51 | 46 | 52 | 58 | 55 | 262

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the End of the Double-blind Treatment in the BPRS (Brief Psychiatric Rating Scale)Total Score
Description: The BPRS consists of 18 ordered categorical items (from "not present" to "extremely severe," on a 1- to 7-point scale), each developed to assess patient symptomatology in a relatively discrete symptom area. The BPRS will be extracted from the PANSS by adding the scores of the 18 items (P2 to P7, N1, N2, and G1 to G10) of the PANSS and will not be assessed separately. The minimum score on the BPRS is 18 and the maximum is 126. The higher number indicates a worsening of schizophrenia.
Time Frame: Baseline and 6 weeks
Population: Intent-to-Treat Division of Neuropharmacological Drug Products Last Observation Carried Forward (ITT-DNDP-LOCF). The ITT-DNDP-LOCF population will include all randomized patients who received at least one dose of study medication and who had at least one efficacy evaluation at Day 3 or beyond, during the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- 40 mg: Lurasidone 40 mg oral tablet taken once a day
- 10 mg Haloperidol: 10 mg Haloperidol overencapsulated tablet taken orally once a day
Arm/Group | 20 mg | 40 mg | 80 mg | 10 mg Haloperidol | Placebo
Number analyzed (Participants) | 71 | 65 | 70 | 72 | 71
units on a scale | -5.0 (1.38) | -5.2 (1.44) | -8.0 (1.40) | -9.8 (1.37) | -7.9 (1.38)
Statistical Analysis 1: Comparison: 20 mg vs 40 mg vs 80 mg vs 10 mg Haloperidol vs Placebo; Test type: Superiority or Other; p < 0.05, ANCOVA

2. Secondary Outcome: Change From Baseline to the End of the Double-blind Treatment in the PANSS (Positive and Negative Syndrome Scale) Scores
Description: The PANSS Positive and Negative Syndrome Scale)is a 30-item scale that evaluates positive, negative, and other symptoms in patients with schizophrenia. Each item is rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme). Scores range from 30-210 with higher scores representing a worsening of schizophrenia.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 20 mg | 40 mg | 80 mg | 10 mg Haloperidol | Placebo
Number analyzed (Participants) | 71 | 65 | 70 | 72 | 71
units on a scale | -7.1 (2.31) | -7.2 (2.42) | -13.6 (2.34) | -16.0 (2.29) | -12.3 (2.32)
Statistical Analysis 1: Comparison: 20 mg vs 40 mg vs 80 mg vs 10 mg Haloperidol vs Placebo; Test type: Superiority or Other; p < 0.05, ANCOVA

3. Secondary Outcome: Change From Baseline to the End of the Double-blind Treatment in the CGI-S (Clinical Global Impression of Severity) Scores
Description: The CGI Severity (CGI-S) assesses the severity of illness of the patient relative to the particular population on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 20 mg | 40 mg | 80 mg | 10 mg Haloperidol | Placebo
Number analyzed (Participants) | 71 | 64 | 70 | 71 | 71
units on a scale | -0.5 (0.11) | -0.4 (0.12) | -0.8 (0.12) | -0.8 (0.12) | -0.7 (0.11)
Statistical Analysis 1: Comparison: 20 mg vs 40 mg vs 80 mg vs 10 mg Haloperidol vs Placebo; Test type: Superiority or Other; p < 0.05, ANCOVA

4. Secondary Outcome: Change From Baseline to the End of the Double-blind Treatment in the MADRS (Montgomery Asberg-Depression Scale) Scores
Description: The MADRS is a 10-item rating scale that assesses apparent and reported sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty in concentration, and lack of interest. Each item is scored on a 7-point scale with a score of 0 reflecting no symptoms and a score of 6 reflecting symptoms of maximum severity.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | 20 mg | 40 mg | 80 mg | 10 mg Haloperidol | Placebo
Number analyzed (Participants) | 71 | 64 | 70 | 72 | 71
units on scale | -1.3 (0.97) | -1.1 (1.02) | -2.5 (0.98) | -2.7 (0.96) | -1.9 (0.97)
Statistical Analysis 1: Comparison: 20 mg vs 40 mg vs 80 mg vs 10 mg Haloperidol vs Placebo; Test type: Superiority or Other; p < 0.05, ANCOVA

ADVERSE EVENTS:
Arm/Group | 20 mg | 40 mg | 80 mg | 10 mg Haloperidol | Placebo
Serious Adverse Events (participants affected / at risk) | 4/71 | 9/67 | 3/71 | 5/72 | 7/72
Other Adverse Events (participants affected / at risk) | 49/71 | 51/67 | 51/71 | 58/72 | 50/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 mg (N=71) | 40 mg (N=67) | 80 mg (N=71) | 10 mg Haloperidol (N=72) | Placebo (N=72)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Grand Mal Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abnormal Behavior (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 2 (2) | 8 (8) | 2 (2) | 3 (3) | 4 (4)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 mg (N=71) | 40 mg (N=67) | 80 mg (N=71) | 10 mg Haloperidol (N=72) | Placebo (N=72)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 6 (6) | 3 (3) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 8 (8) | 6 (6) | 8 (8) | 5 (5) | 7 (7)
Nausea (Gastrointestinal disorders) | 8 (8) | 7 (7) | 13 (13) | 4 (4) | 8 (8)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Vomiting (Gastrointestinal disorders) | 5 (5) | 5 (5) | 12 (12) | 4 (4) | 5 (5)
Fatigue (General disorders) | 5 (5) | 2 (2) | 9 (9) | 7 (7) | 3 (3)
Pain (General disorders) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 5 (5)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 2 (2) | 4 (4) | 1 (1)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 5 (5) | 4 (4) | 2 (2)
Akathisia (Nervous system disorders) | 4 (4) | 9 (9) | 13 (13) | 14 (14) | 7 (7)
Dizziness (Nervous system disorders) | 4 (4) | 3 (3) | 4 (4) | 3 (3) | 3 (3)
Dystonia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 9 (9) | 1 (1)
Extrapyramidal Disorder (Nervous system disorders) | 3 (3) | 4 (4) | 4 (4) | 13 (13) | 3 (3)
Headache (Nervous system disorders) | 15 (15) | 16 (16) | 17 (17) | 14 (14) | 24 (24)
Sedation (Nervous system disorders) | 8 (8) | 11 (11) | 15 (15) | 15 (15) | 6 (6)
Somnolence (Nervous system disorders) | 3 (3) | 4 (4) | 7 (7) | 9 (9) | 4 (4)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 1 (1)
Agitation (Psychiatric disorders) | 7 (7) | 9 (9) | 3 (3) | 3 (3) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2) | 9 (9) | 2 (2) | 9 (9) | 4 (4)
Insomnia (Psychiatric disorders) | 6 (6) | 5 (5) | 4 (4) | 12 (12) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 1 (1) | 1 (1) | 5 (5)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 2 (2) | 2 (2) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 2 (2) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No